CLINICAL TRIAL: NCT01601743
Title: Exercise as a Behavioral Treatment for Cocaine Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Richard De La Garza, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-27380; 1R21DA030722 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2012-02-20; First posted 2012-05-18 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2012-05

CONDITIONS: Cocaine Dependence; Cocaine Addiction; Cocaine Abuse; Substance Abuse
Keywords: Cocaine; Exercise
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders; Motor Activity | interventions — Sitting Position; Running; Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sitting (Active Comparator): Sitting for the same period of time and duration (30 minutes per session, 3 times per week, over 4 consecutive weeks).
  Interventions: Behavioral: Sitting
- Running (Active Comparator): Exercise (running) for 30 minutes per session, 3 times per week, over 4 consecutive weeks.
  Interventions: Behavioral: Running
- Walking (Active Comparator): Exercise (walking) for 30 minutes per session, 3 times per week, over 4 consecutive weeks.
  Interventions: Behavioral: Walking

INTERVENTIONS:
Behavioral: Sitting — Sitting for the same period of time and duration (30 minutes per session, 3 times per week, over 4 consecutive weeks).
  Arms: Sitting
Behavioral: Running — Exercise (running) for 30 minutes per session, 3 times per week, over 4 consecutive weeks.
  Arms: Running
Behavioral: Walking — Exercise (walking) for 30 minutes per session, 3 times per week, over 4 consecutive weeks.
  Arms: Walking

SUMMARY:
The purpose of this study is to test the effects of exercise on cocaine use, fitness, and cravings for cocaine and nicotine. This study is part of an effort to develop treatments for cocaine abuse.

DETAILED DESCRIPTION:
This proposal represents an important research effort with considerable public health significance in that it will provide detailed behavioral and physiological data for a non-pharmacological intervention to treat stimulant addiction. Regular exercise is known to promote better mental and physical health, however the effects of exercise on cocaine use and craving in cocaine-dependent individuals has not been previously assessed. The Specific Aims include: 1) To evaluate the effects of regular exercise (running and walking) versus placebo (sitting) on basic fitness measures; 2) To evaluate the effects of exercise on objective and subjective measures of cocaine and nicotine use and craving. Participants will also receive a total of 12 sessions of a standardized series of computerized cognitive behavioral therapy (CCBT) modules, which are specifically designed for the treatment of cocaine addiction.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in the study, participants must:

* 1. Be English-speaking volunteers between 21-55 years of age
* 2. Be cocaine-dependent and nicotine-dependent (>10 cigarettes/day and FTND >4)
* 3. Be seeking treatment for cocaine dependence
* 4. Have vital signs as follows: resting pulse between 50-90 bpm, supine blood pressures between 85-150 mmHg systolic and 45-90 mmHg diastolic
* 5. Have a breathalyzer test indicating an undetectable blood alcohol level
* 6. Have a medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician and the PI. Most relevant, assessments will include the participants' general health and suitability for inclusion in a rigorous exercise program.

Exclusion Criteria:

Potential participants will be excluded if any of the following apply:

* 1. Have neurological or psychiatric disorders, as assessed by MINI, such as: a. current major depression; b. lifetime history of schizophrenia, other psychotic illness, or bipolar illness; c. current organic brain disease or dementia assessed by clinical interview; d. current psychiatric disorder as assessed by the MINI including history of suicide attempts within the past three months and/or current suicidal ideation/plan
* 2. Meet DSM-IV criteria for abuse or dependence on other drugs, except for cocaine or nicotine
* 3. Have any of the conditions defined by the American College of Sports Medicine (2006) as "absolute contraindications to exercise testing"
* 4. Have evidence of clinically significant heart disease or hypertension
* 5. Have evidence of clinically significant or unstable medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease
* 6. Be pregnant or nursing. All females must provide a negative pregnancy urine test
* 7. Currently use alpha or beta agonists, theophylline, or other sympathomimetics
* 8. Currently engaged in an exercise regimen of similar intensity as those planned for investigation
* 9. Have any other illness, condition, or use of medications, which in the opinion of the PI and/or the study physician would preclude safe and/or successful completion of study.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The effects of exercise on cardiovascular and basic fitness measures | 4 weeks
  Before and after each exercise session, physiologic responses will be closely monitored using repeated HR, BP, and ECG readings. To evaluate safety, a DSMB will meet annually and following any serious AE to examine data as well as any new published information on exercise relevant to the project. The number of AEs (including arrhythmias and ECG changes), changes in BP and HR, and changes in mood and psychiatric symptoms (using the BSI, BDI, POMS, and BPRS) will also be assessed throughout the study.

SECONDARY OUTCOMES:
The effects of exercise on changes in drug use measures and in self-reported craving for cocaine and/or nicotine | 4 weeks
  The effects of exercise (running vs. walking 30 min per session, 3 times per week, over 4 consecutive weeks) versus placebo (sitting for the same period of time and duration) on self-reports of craving for cocaine/nicotine will be measured by the Brief Substance Craving Scale (BSCS), Wisconsin Smoking Withdrawal Scale (WSWS), and the Questionnaire of Smoking Urges (QSU-Brief) throughout the 4-week study period and at 2 follow-up visits.
The effects of exercise on Brain Derived Neurotrophic Factor (BDNF) in blood samples | 4 weeks
  The effects of exercise versus placebo on changes in BDNF will be measured, since exercise has been shown to increase BDNF and neurogenesis in the hippocampus. Approximately 2 mls of blood will be taken for BDNF analysis at six timepointss during and after the study: 1) On day 1 prior to randomization 2) once weekly on Fridays - i.e., 4 measures at end of treatment at Week 1, 2, 3, and 4. Samples will be taken 20 minutes before participants run, walk or sit. 3) at follow up visit (39 weeks or 52 weeks).
The effects of exercise on changes in drug use measures | 4 weeks
  The effects of exercise (running vs. walking 30 min per session, 3 times per week, over 4 consecutive weeks) versus placebo (sitting for the same period of time and duration) on changes in drug use will be assessed by measuring urine toxicology and salivary nicotine and cotinine throughout the 4-week study and at 2 follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Richard De La Garza, II, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas, United States